CLINICAL TRIAL: NCT03073577
Title: Clinical Study Using Antiaging Glycopeptide (PKX-001) in Islet Transplantation
Brief Title: Islet Transplantation Using PKX-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: ProtoKinetix Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00067564
Record Dates: First submitted 2017-02-26; First posted 2017-03-08 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Islet Transplantation; Diabetes; Diabetes Treatment
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — AAGP glycopeptide, 580 Da

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): PKX-001 will be supplemented to islet preservation CMRL-1066 medium at final concentration of 3 mg/mL during islet isolation process. On the day of transplantation, preserved islets supplemented with PKX-001 are collected and washed with Transplant Media, which does not contain PKX-001, as a standard procedure. The isolation team will evaluate the final islet product based on standard assays. Islets are maintained for minimal 6 hours up to 72 hours in supplemented CMRL1066-based media containing PKX-001 until the time of transplant. When product release minimal criteria are met, islets will be clinically transplanted into patients intraportally.
  Interventions: Drug: Antiaging Glycopeptide

INTERVENTIONS:
Drug: Antiaging Glycopeptide — Antiaging Glycopeptide (PKX-001) will be supplemented to islet preservation medium during islet isolation process. On the day of transplantation, preserved islets supplemented with PKX-001 are collected and washed with Transplant Media, which does not contain PKX-001, as a standard procedure. The isolation team will evaluate the final islet product based on standard assays used in standard of care practice. When product release minimal criteria are met, islets will be clinically transplanted into patients intraportally by percutaneous transhepatic access.
  Other Names: PKX-001; AAGP

SUMMARY:
Islet Transplantation is a procedure used in people with difficult to control Type 1 Diabetes. Insulin producing cells (islets) are isolated from a deceased donor pancreas. After the cells are carefully isolated from the donor pancreas, the islets are transplanted into the recipient's liver. These transplanted islets may produce insulin.

One of the challenges with islet transplant is the death of some of the transplanted islets due to inflammation, oxidative stress and exposure to diabetogenic immunosuppressive agents associated with islet functional impairment and graft loss, especially linked to the use of calcineurin inhibitors, including tacrolimus (Tac).

Antiaging glycopeptide (PKX-001) is a small, stable, synthetic replica of antifreeze proteins (AFPs), which naturally occur in Arctic and Antarctic fish and have been shown protecting cells against harmful conditions. PKX-001 is a new drug that has been shown in lab studies to help islet cells survive isolation and keep them healthy and functioning. Most importantly, animal studies have shown that islets treated with PKX-001 were protected from the immunosuppressant (Tac) toxicity and retained their function in animals receiving islet transplant.

This study will involve up to 10 participants from the islet transplant waiting list at the Clinical Islet Transplant Program. All participants will receive islets treated with the medication PKX-001. PKX-001 will be used only in the islet preservation process, and will not be given to participants as medication.

The purpose of this study is to confirm the safety of transplantation of PKX-001 treated islets and to evaluate the cytoprotective capacity of PKX-001 in islet transplantation, especially its capacity to protect against Tac induced graft dysfunction.

DETAILED DESCRIPTION:
Background

Clinical islet transplantation is today an accepted modality to treat selected diabetic patients with frequent hypoglycemic events and severe glycemic liability. Although islet transplantation outcomes have improved significantly in highly specialized centers with a 5-year insulin independence rate exceeding 50%, a proportion of patients require reintroduction of insulin later on. Tac may be partly responsible for the limited islet durability and the need for multiple donors for each recipient in spite of its ability to prevent rejection and autoimmune recurrence. In vitro studies of islets exposed to immunosuppressants have shown that Tac levels above 10-100 mg/L cause vacuolization and destruction of islets in culture.

Antifreeze proteins (AFPs) have generated considerable interest for their ability to protect cells under a variety of conditions. However, their large size restricts their use in medicine as they are unable to pass through capillaries into interstitial tissue and are unable to reach target cells.

With these disadvantages of AFPs in mind, Dr. Geraldine-Castelot-Deliencourt (Rouen, France) invented Antiaging glycopeptide, which is later manufactured by ProtoKinetix Inc. (St. Marys, West Virginia, US). ProtoKinetix' anti-aging glycopeptide, PKX-001, is a small, stable, synthetic replica of the larger, less stable AFP.

PKX-001 has gone through a series of tests in various outsourced laboratories in Europe and North America. These tests have proven its ability to protect a multitude of cell lines (Hela cells, adult fibroblast, neonatal fibroblasts, human neuronal stem cells, mouse neuronal stem cells, mouse islet cells, blood platelets, cluster of differentiation 34+ (CD34+) cells, and keratinocytes) against ultraviolet A (UVA), ultraviolet C (UVC), Hydrogen Peroxide, Inflammatory (ILβ), Time, Temperature (-196°C, -80°C, -3°C, 3°C, 4°C, 15°C and 22°C) and Low Serum induced cell death at pHs from 5.3 -10.5. In addition to protecting cell survival PKX-001 also preserves cell functionality. This has been tested via stem cell markers, CD34+ functionality tests, and in vivo studies where PKX-001 treated transplanted islet cells were found to reduce blood glucose concentrations in diabetic mice by 40% by day 40 in comparison to islet cells which were transplanted into mice without first being exposed to PKX-001.

In light of the beneficial roles of PKX-001 on cellular survival and functionality preservation, our team have evaluated the cytoprotective capacity of PKX-001 in islet transplant, especially its capacity of protection against the diabetogenic effect of Tac.

In vitro assessment of human islets in culture with PKX-001 supplementation has also showed enhanced quality and yield of post-preservation human islets and protection against acute exposure to Tac at clinical relevant doses compared with those without PKX-001 supplementation. Further analysis indicated that islets treated with PKX-001 had decreased oxidative stress, improved insulin release by increasing islet exocytosis, decreased islet loss during preservation due to apoptosis, even in the presence of Tac.

In vivo studies have complemented all in vitro findings above, which demonstrated that PKX-001 supplementation suppressed early inflammation and improved islet engraftment with long-term efficacy.

The proposed study is a phase I, non-randomized, open-label, single arm, prospective trial using retrospective controls.

Ten adult Islet transplant candidates (18 years and older), deemed appropriate for standard islet transplant at the University of Alberta Hospital will be enrolled in this investigation.

Retrospective data from 10 islet transplant patients consented for chart review (Protocol #: 000001120 entitled: "On-going review of islet transplant patients at the University of Alberta" and Protocol #: 000001122 entitled: "Collaborative Islet Transplant Registry") will be also collected.

The standard of Care controls will be identified from the Islet Transplant program database (period: 2014 - 2016) and anonymized by a simple numbering system.

Hypothesis:

Transplantation of PKX-001 treated islets is safe and improves graft outcomes.

Primary Objective:

To demonstrate safety of transplantation of PKX-001 treated islets.

Secondary Objectives:

To assess efficacy of transplantation of PKX-001 treated islets To assess efficacy of addition of PKX-001 during islet preservation

Procedures:

Prior to transplantation, the patient is screened, qualified, listed for transplant, and signs the informed consent form.

At the time a suitable islet preparation becomes available, the patient will receive allogeneic islet cells transplanted into patients intraportally by percutaneous transhepatic access.

Islet transplant will be performed under the current immunosuppression regimen including: induction (Alemtuzumab/Basiliximab) and long-term immunosuppression (Prograf/Cellcept). The engraftment regimen includes anti-inflammatory medications (Etanercept/Anakinra) and intravenous insulin and heparin. The only additional intervention used in this pilot trial is the addition of the investigational agent, PKX-001 to islet processing.

Follow up:

Participants will undergo a 3-month follow-up period following their initial or subsequent islet transplant.

There are no study-specific follow-up visits required for this study. Study subjects will be followed as per standard of care. For the purpose of evaluating the primary and secondary endpoints, the following measurements collected on study subjects at the time points indicated as per standard of care, will be chart reviewed and recorded up to Day 30 post-transplant:

Clinical Assessment by Transplant Fellow or Staff; Post-Transplant Blood work (as per Standard of Care); Metabolic testing: Ensure (or Arginine); Glucose Records for Self-Monitoring. Incidence of Primary Non-Function (see Glossary for definition); Incidence of Adverse Events or Serious Adverse Events can be reported on any day post transplant; Abdominal Ultrasound with Doppler report (clinically significant findings). The study will remain open to collect all 10 recipients' follow-up data to 3 month post-transplant. Primary and secondary outcome reporting will occur 90 days following the transplant of the last patient to the trial.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible the participant must have had type 1 diabetes mellitus (T1DM) for more than 5 years, complicated by at least 1 of the following situations that persist despite intensive insulin management efforts:

  1. Reduced awareness of hypoglycemia, as defined by the absence of adequate autonomic symptoms at plasma glucose levels < 3.0 mmol/L, indicated by, 1 or more episodes of severe hypoglycemia requiring third party assistance within 12 months, a Clarke score ≥4, hypoglycemic (HYPO) score ≥1,000, lability index (LI) ≥400 or combined HYPO/LI >400/>300.
  2. Metabolic instability, characterized by erratic blood glucose levels that interfere with daily activities and/or 1 or more hospital visits for diabetic ketoacidosis over the last 12 months.

     Participants must be capable of understanding the purpose and risks of the study and must sign a statement of informed consent.
* Retrospective Control Inclusion Criteria:

All control participants will be included according to the immunosuppression / engraftment regimen used in this pilot, specifically the current standard of care islet transplant at the University of Alberta Hospital: Alemtuzumab/Basiliximab, Anakinra, Etanercept, Mycophenolate Mofetil and Tacrolimus.

Exclusion Criteria:

* History of enrollment in any other islet transplant trials (at the discretion of the investigator).
* Severe co-existing cardiac disease, characterized by any one of these conditions: (a) recent (within the past 6months) myocardial infarction; (b) left ventricular ejection fraction <30%; or (c) evidence of ischemia on functional cardiac exam.
* Active alcohol or substance abuse, to include cigarette smoking (must be abstinent for 6 months prior to listing for transplant).
* Psychiatric disorder making the patient not a suitable candidate for transplantation (e.g., schizophrenia, bipolar disorder, or major depression that is unstable or uncontrolled on current medication).
* History of non-adherence to prescribed regimens.
* Active infection including Hepatitis C, Hepatitis B, HIV, or Tuberculosis (TB) (subjects with a positive purified protein derivative (PPD) performed within one year of enrollment, and no history of adequate chemoprophylaxis).
* Any history of, or current malignancies except squamous or basal skin cancer.
* BMI > 35 kg/m2 at screening visit.
* Age less than 18 or greater than 68 years.
* Measured glomerular filtration rate (GFR) <60 mL/min/1.73 m2.
* Presence or history of macroalbuminuria (>300 mg/g creatinine).
* Clinical suspicion of nephritic (hematuria, active urinary sediment) or rapidly progressing renal impairment (e.g. Increase in serum creatinine of 25% within the last 3-6 months).
* Baseline Hb < 105g/L (<10.5 g/dL) in women, or < 120 g/L (<12 g/dL) in men.
* Baseline screening liver function tests outside of normal range, with the exception of uncomplicated Gilbert's Syndrome. An initial liver function test (LFT) panel with any values >1.5 times the upper limit of normal (ULN) will exclude a patient without a re-test; a re-test for any values between ULN and 1.5 times ULN should be made, and if the values remain elevated above normal limits, the patient will be excluded.
* Untreated proliferative retinopathy.
* Positive pregnancy test, intent for future pregnancy or male subjects' intent to procreate, failure to follow effective contraceptive measures, or presently breast-feeding.
* Evidence of significant sensitization on panel reactive antibody (PRA) (at the discretion of the investigator).
* Insulin requirement >1.0 U/kg/day
* HbA1C >12%.
* Uncontrolled hyperlipidemia [fasting LDL cholesterol > 3.4 mmol/L (133 mg/dL), treated or untreated; and/or fasting triglycerides > 2.3 mmol/L (90 mg/dL)].
* Under treatment for a medical condition requiring chronic use of steroids.
* Use of coumadin or other anticoagulant therapy (except aspirin) or patient with prothrombin time (PT) / international normalized ratio (INR) > 1.5.
* Untreated Celiac disease.
* Patients with Graves disease will be excluded unless previously adequately treated with radioiodine ablative therapy.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Adverse event morbidity | Up to 1 year post-transplant
  Adverse event morbidity within 1 year post-transplant
Serious adverse event morbidity | Up to 1 year post-transplant
  Adverse event morbidity within 1 year post-transplant

SECONDARY OUTCOMES:
Number of participants with insulin independence | Day 90 post-transplant
  Number of participants who achieve insulin independence at Day 90 post-transplant
Islet yield | Day 0
  Difference in islet yield between treatment group and current standard protocol data
Engraftment index | Day 90 post-transplant
  Difference in engraftment index between treatment group and current standard protocol data
Islet viability | Day 0
  Difference in islet viability between treatment group and current standard protocol data
Glucose stimulated insulin release | Day 0
  Difference in glucose stimulated insulin release between treatment group and current standard protocol data
Oxygen consumption ratio | Day 0
  Difference in oxygen consumption ratio between treatment group and current standard protocol data
Insulin requirement | Day 0
  Difference in insulin requirement between treatment group and current standard protocol data
Beta-2 score | Day 0
  Difference in beta-2 score between treatment group and current standard protocol data

CONTACTS AND LOCATIONS:
Overall Officials: James Shapiro, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: related information — http://www.islet.ca/